CLINICAL TRIAL: NCT01610596
Title: A Double-blind, Randomized, Multicenter, Vehicle-Controlled Parallel Group Study to Determine the Efficacy and Safety of Halobetasol Propionate Lotion 0.05% in Subjects With Plaque Psoriasis Receiving Two Weeks of Treatment
Brief Title: A Study to Determine the Efficacy and Safety of Halobetasol Propionate Lotion 0.05% in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000-0551-207
Record Dates: First submitted 2012-01-18; First posted 2012-06-04 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: Psoriasis; Skin Diseases; Halobetasol; Vasoconstrictor Agents; Therapeutic Uses; Pharmacologic Actions; Anti-Inflammatory Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Halobetasol Propionate Lotion 0.05% (Experimental): Topical lotion, applied twice daily
  Interventions: Drug: Halobetasol Propionate Lotion 0.05%
- Vehicle Lotion (Placebo Comparator): Topical lotion, applied twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Halobetasol Propionate Lotion 0.05% — Apply twice daily for 1-2 weeks, not to exceed 50 grams per week
  Arms: Halobetasol Propionate Lotion 0.05%
Drug: Placebo
  Arms: Vehicle Lotion

SUMMARY:
This is a double-blind, multicenter, vehicle-controlled, parallel group comparison study to determine and compare the efficacy and safety of HBP Lotion 0.05% and Vehicle Lotion applied twice daily for two weeks in subjects with moderate to severe plaque psoriasis. Eligible subjects will be randomized (1:1) to one of two treatment groups - HBP Lotion 0.05% or Vehicle Lotion. The maximum amount of test article to be applied per week should not exceed 50 grams.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is Male or non-pregnant female; 18 years of age at time of Screening.
2. Subject is willing and able to give written informed consent.
3. subject is willing and able to apply the test article(s) as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
4. Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than approximately 10% body surface area (BSA) (excluding the face, scalp, groin, axillae and other intertriginous areas).
5. Subject has an Overall Disease Severity (ODS) score for the Treatment Area of at least three (3) at the Baseline Visit.
6. If subject is a woman of childbearing potential (WOCBP) , she must have a negative urine pregnancy test (UPT) and agree to use an effective form of birth control for the duration of the study (i.e., abstinence, stabilized on hormonal contraceptives [oral, injectable, transdermal or intravaginal] or IUD for at least three months prior to test article application, condom and a spermicidal, or diaphragm and a spermicidal). Abstinence is an acceptable form of birth control for subjects who are not sexually active. Subjects who become sexually active during the trial must agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
3. Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, or which exposes the subject to an unacceptable risk by study participation.
4. Subject has used any phototherapy (including laser), photo-chemotherapy or systemic corticosteroid therapy (such as systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids]) within 30 days prior to the Baseline Visit.
5. Subject has used any systemic methotrexate, retinoids, cyclosporine or analogous products within 90 days prior to the Baseline Visit.
6. Subject has used any systemic biologic therapy (i.e., FDA approved or experimental therapy) within five (5) half-lives of the biologic prior to the Baseline Visit. Published or documented half-life of the product provided by the commercial supplier or Sponsor should be used to establish this value.
7. Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the Baseline Visit or is intending to have such exposure during the study that is thought by the investigator likely to modify the subject's disease.
8. Subject has used topical body (excluding the scalp) psoriasis therapy including coal tar, anthralin, steroids, retinoids, vitamin D analogs (e.g., Dovonex®) within 14 days prior to the Baseline Visit.
9. Subject has used emollients/moisturizers on areas to be treated within four hours prior to clinical evaluation at the Baseline Visit.
10. Subject is currently using lithium or Plaquenil (hydroxychloroquine).
11. Subject is currently using a beta-blocking medication (e.g., propanolol) or angiotensin converting enzyme (ACE) inhibitor at a dose that has not been stabilized, in the opinion of the investigator.
12. Subject has a history of sensitivity to any of the ingredients in the test article.
13. Subject is pregnant, lactating, or is planning to become pregnant during the study.
14. Subject is currently enrolled in an investigational drug or device study.
15. Subject has used an investigational drug or investigational device treatment within 30 days prior to the Baseline Visit.
16. Subject has been previously enrolled in this study and treated with a test article.
17. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, PhD, Study Director — Therapeutics, Inc.
Locations (3):
- United States (3):
  - Therapeutics Clinical Research, San Diego, California
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - DermResearch, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2011 to February 2012
  The location of clinical sites included dermatology clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Groups:
- Halobetasol Propionate Lotion 0.05%: Topical lotion, applied twice daily
  Halobetasol Propionate Lotion 0.05%: Apply twice daily for 2 weeks, not to exceed 50 grams per week
- Vehicle Lotion: Topical lotion, applied twice daily
  Placebo
Period: Overall Study
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Started | 36 | 36
Completed | 36 | 35
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analyses are based on the Safety population. All participants enrolled in the study who were dispensed and applied test article at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (11.74) | 52.3 (13.06) | 51.2 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 28 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 25 | 33 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 32 | 34 | 66
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Overall Disease Severity at Baseline [Number; unit: participants] — To be enrolled into the study, subjects had to have at least moderate ODS (score of at least 3). One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 30 | 31 | 61
    Severe/very severe | 6 | 5 | 11
Signs of Psoriasis at Baseline (scaling) [Number; unit: participants] — One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 6 | 2 | 8
    Moderate | 22 | 28 | 50
    Severe/very severe | 8 | 6 | 14
Signs of Psoriasis at Baseline (erythema) [Number; unit: participants] — One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  participants
    Clear | 0 | 0 | 0
    Almost clear | 1 | 0 | 1
    Mild | 1 | 1 | 2
    Moderate | 22 | 24 | 46
    Severe/very severe | 12 | 11 | 23
Signs of Psoriasis at Baseline (plaque elevation) [Number; unit: participants] — One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 2 | 3 | 5
    Moderate | 30 | 28 | 58
    Severe/very severe | 4 | 5 | 9
Pruritus at Baseline [Number; unit: participants] — This evaluation is the participant's assessment of the itch on the active psoriasis plaques based on the 5-point Itch Evaluation Scoring Scale Form. One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  participants
    None | 3 | 8 | 11
    Mild | 14 | 5 | 19
    Mild to moderate | 12 | 11 | 23
    Moderate | 5 | 5 | 10
    Moderal to severe | 1 | 5 | 6
    Severe | 1 | 2 | 3
Percent BSA to be Treated at Baseline [Mean (Standard Deviation); unit: %BSA] — The percent Body Surface Area (BSA) with active psoriasis within the designated Treatment Area was assessed at Baseline. One study participant (vehicle group) did not return to the clinic (lost to follow-up) following Visit 1 (baseline visit) and was therefore excluded from the Intent-to-Treat (ITT) population.
  %BSA | 3.7 (1.74) | 4.0 (2.04) | 3.8 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease Severity Score (Success)
Description: Overall disease severity (ODS) will be recorded at baseline, Day 8, and Day 15 on a 0 (clear) to 4 (severe/very severe) point scale. The primary efficacy endpoint was the percentage of subjects with ODS treatment "success" at end of treatment (Day 15). Success was defined as a grade of 0 or 1 on the ODS scale.
Time Frame: Day 15
Population: Analysis shown is the Intent-to-treat (ITT) population, defined as all enrolled participants who were randomized and applied at least one dose of the test article.
Measure: Number; unit: percentage of participants
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Number analyzed (Participants) | 36 | 35
percentage of participants | 30.6 | 0.0
Statistical Analysis 1: Comparison: Halobetasol Propionate Lotion 0.05% vs Vehicle Lotion; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Percent Body Surface Area
Description: Changes in percent BSA with active psoriasis in the Treatment Area
Time Frame: Baseline, Days 8 and 15
Population: Analysis shown is based on the ITT population.
Measure: Mean (Standard Deviation); unit: Change in %BSA
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Number analyzed (Participants) | 36 | 35
Change in %BSA
  at Day 8 | -0.3 (0.57) | -0.1 (0.34)
  at Day 15 | -1.3 (1.34) | -0.2 (0.93)

3. Secondary Outcome: Clinical Signs and Symptoms of Psoriasis
Description: The proportion of subjects rated a "treatment success" for each of the clinical signs and symptoms of psoriasis: scaling, erythema, plaque elevation and pruritis. "Treatment success" is defined as a score of 0 or 1 on a five-point scale ranging from 0 = clear to 4 = severe/very severe.
Time Frame: Days 8 and 15
Population: Analysis shown is based on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Number analyzed (Participants) | 36 | 35
percentage of participants
  Scaling (Day 8) | 25.0 | 8.6
  Scaling (Day 15) | 61.1 | 11.4
  Erythema (Day 8) | 2.9 | 0.0
  Erythema (Day 15) | 13.9 | 2.9
  Plaque elevation (Day 8) | 11.1 | 0.0
  Plaque elevation (Day 15) | 38.9 | 2.9

4. Secondary Outcome: Overall Disease Severity Score (Improvement)
Description: The proportion of subjects rated a "improved" for ODS at Day 8 and Day 15. "Improvement" is defined as at least a two (2) grade decrease in severity score relative to baseline using a five-point scale ranging from 0 = clear to 4 = severe/very severe.
Time Frame: Days 8 and 15
Measure: Number; unit: percentage of participants
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Number analyzed (Participants) | 36 | 35
percentage of participants
  at Day 8 | 13.9 | 0.0
  at Day 15 | 44.4 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 15) or early participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The Safety population included all participants enrolled in the study who were dispensed the test article at least once; all participants enrolled in the study applied the first application in the clinic and were included in the Safety population.
Arm/Group | Halobetasol Propionate Lotion 0.05% | Vehicle Lotion
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 11/36 | 5/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Halobetasol Propionate Lotion 0.05% (N=36) | Vehicle Lotion (N=36)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site atrophy (General disorders) | 2 (2) | 0 (0)
Application site discoloration (General disorders) | 1 (2) | 0 (0)
Application site pain (General disorders) | 3 (3) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.